CLINICAL TRIAL: NCT01094808
Title: Effect of Pregabalin on Colonic Sensorimotor Function in Healthy Adults.
Brief Title: Pregabalin and Colonic Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Michael Camilleri, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 09-008469; 1RC1DK086182 (NIH); R01DK079866 (NIH); R01DK067071 (NIH); UL1RR024150 (NIH)
Record Dates: First submitted 2010-03-24; First posted 2010-03-29 (Estimated); Results first posted 2012-03-06 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
Keywords: pregabalin; motor; sensation; colon; pain; gas
MeSH Terms: conditions — Pain; Mucopolysaccharidosis IV | interventions — Pregabalin; Cathartics; Golytely

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pregabalin 75 mg (Experimental): Subjects randomized to this arm received a single dose of pregabalin 75 mg orally
  Interventions: Drug: Pregabalin; Other: Bowel preparation
- Pregabalin 200 mg (Experimental): Subjects randomized to this arm received a single dose of pregabalin 200 mg orally
  Interventions: Drug: Pregabalin; Other: Bowel preparation
- Placebo (Placebo Comparator): Subjects randomized to this arm received a single dose of placebo medication orally
  Interventions: Drug: Placebo; Other: Bowel preparation

INTERVENTIONS:
Drug: Pregabalin — FDA approved medication (capsules) at 75 mg and 200 mg doses
  Other Names: Lyrica
  Arms: Pregabalin 200 mg; Pregabalin 75 mg
Drug: Placebo — Placebo capsules
  Arms: Placebo
Other: Bowel preparation — Polyethylene glycol electrolyte solution bowel preparation
  Other Names: GoLYTELY

SUMMARY:
This study is being done to evaluate the effects of pregabalin, a drug approved for anticonvulsive therapy and for neuropathic pain, on colonic and sensory functions in healthy individuals.

The specific study hypotheses were as follows: 1) pregabalin increases sensation thresholds, decreases sensation ratings, and increases compliance in response to balloon distension in the colon; 2) pregabalin reduces colonic phasic and tonic motility in response to a standardized meal; and 3) sensation ratings are lower with higher colonic compliance.

DETAILED DESCRIPTION:
The treatment of patients with irritable bowel syndrome and chronic abdominal pain is advancing with several effective options for symptoms related to bowel dysfunction and bloating/distension. However, there are no approved or effective centrally or peripherally acting visceral analgesics. Pregabalin has been proposed as a treatment for visceral pain, based on the pharmacological actions, and efficacy in neuropathic pain.

This was a trial of healthy adults to compare the effects of oral pregabalin, 75 mg and 200 mg versus placebo on sensation and contraction of the colon using validated methods.

All participants presented on the study day after an overnight bowel preparation with an oral colonic lavage solution and a 12-hour fast. Flexible colonoscopy to the splenic flexure was performed without sedation by one investigator. The barostat catheter (constructed at Mayo Clinic, Rochester, MN) incorporating six manometric point sensors 5 cm apart was introduced into the colon over a guidewire, and the polyethylene balloon (10 cm long, cylindrical shape with a maximum volume of 600 ml) was placed in the mid-descending or junction of the sigmoid and descending colon. A rigid-piston barostat was used to measure intraballoon pressure and volume throughout the study. After an initial inflation to a volume of 75 ml to ensure unfolding of the balloon, the operating pressure was identified as the distension pressure at which respiratory excursions were recorded clearly from the barostat tracing, and the intraballoon pressure was set 2 mm Hg above the minimal distension pressure. A conditioning distention from 0 to 36 mm Hg in increments of 4 mm Hg every 15 seconds was performed over a period of 3 minutes.

After an equilibration period of 10 minutes, colonic compliance was assessed by the ascending methods of limit (ramp-like increases of 4 mm Hg at 30 section intervals). During the assessment of colonic compliance, participants reported their thresholds for first perception, gas and pain. After another 10 minute equilibration period, fasting colonic tone was measured at operating pressure for a period of 10 minutes.

Randomized-order phasic distentions were then applied at 16, 24, 30, and 36 mm Hg above the operating pressure to measure the sensations of gas and pain. Each distention lasted 1 minute and was followed by an equilibration period at the operating pressure for 2 minutes. A 100-mm visual analog scale (VAS) was used to assess the rating of arousal and stress experienced by each participant before performing the phasic distentions. During the distentions, participants also used the 100-mm VAS to rate the intensity of gas and pain perception at 30 seconds from the start of the distention.

Colonic compliance, fasting tone, pressure thresholds for first perception, gas, and pain, and VAS scores of gas and pain during the phasic distentions were measured before administering the study medication and 1 hour after drug administration. After the postdrug assessment of sensation with phasic distentions, a 30-min assessment of fasting colonic tone was measured in each participant; this provided a baseline to compare the effect of a standard 750-ml chocolate milkshake meal across treatment groups. Postprandial tone was measured over 60 minutes, with the main focus on the first 30 minutes. When the recording was completed, the balloon was deflated and the tube removed by gentle traction.

ELIGIBILITY:
Inclusion criteria:

- Healthy males or females

Exclusion criteria:

* Abdominal surgery other than appendectomy, laparoscopic cholecystectomy, cesarean section, vaginal or laparoscopic hysterectomy or tubal ligation
* A history of chronic gastrointestinal or systemic illnesses that could affect gastrointestinal motility
* Any history of hypertension
* Use of medications that may alter gastrointestinal motility or interact with the study medications
* Use of any of the study medications within the past 30 days
* Pregnancy
* Chronic renal insufficiency (serum creatinine >1.5 mg/dL)
* Psychiatric or psychologic dysfunction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Iturrino J, Camilleri M, Busciglio I, Burton D, Zinsmeister AR. Effect of the alpha2delta ligand, pregabalin, on colonic sensory and motor functions in healthy adults. Am J Physiol Gastrointest Liver Physiol. 2011 Aug;301(2):G377-84. doi: 10.1152/ajpgi.00085.2011. Epub 2011 May 19. PMID 21596994
- [Derived] Iturrino J, Camilleri M, Busciglio I, Burton D, Zinsmeister AR. Sensations of gas and pain and their relationship with compliance during distension in human colon. Neurogastroenterol Motil. 2012 Jul;24(7):646-51, e275. doi: 10.1111/j.1365-2982.2012.01901.x. Epub 2012 Mar 6. PMID 22393902

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between April 2010 and January 2011 at the Mayo Clinic, Rochester, Minnesota.
Period: Overall Study
Arm/Group | Pregabalin 75 mg | Pregabalin 200 mg | Placebo
Started | 21 | 20 | 21
Completed | 20 | 19 | 21
Not Completed | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin 75 mg | Pregabalin 200 mg | Placebo | Total
Number analyzed (Participants) | 21 | 20 | 21 | 62
Age Continuous [Mean (Standard Deviation); unit: years] | 32.2 (11.9) | 32.4 (9.1) | 31.6 (11.8) | 32 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 15 | 46
  Male | 5 | 5 | 6 | 16
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 21 | 62
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body mass index is defined as the individual's body weight divided by the square of his or her height.
  kg/m^2 | 25.8 (3.7) | 26.7 (6.3) | 26.4 (4.4) | 26.3 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Sensory Threshold for Pain
Description: The sensory threshold for first perception of pain was measured by stepwise inflation of the balloon in increments of 4 mm Hg at 60 second intervals. The balloon was placed in the mid-descending or junction of the sigmoid and descending colon. During this assessment participants were asked to report when they had the first perception of pain. The investigator recorded the threshold pressure at which the participants reported this sensation.
Time Frame: approximately 60 minutes after drug administration
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Pregabalin 75 mg | Pregabalin 200 mg | Placebo
Number analyzed (Participants) | 20 | 19 | 21
mm Hg | 45.8 (14.9) | 46.7 (13.9) | 45.0 (14.0)

2. Primary Outcome: Sensation Ratings for Pain and Gas at 30 mm Hg Distension Above Baseline Operating Pressure
Description: The 30 mm Hg distension refers to inflation of the balloon placed in placed in the mid-descending or junction of the sigmoid and descending colon. Pain and gas were individually measured by a 100 mm long Visual Analog Scale (VAS). The VAS does not have any pre-set marks between the extremes. For the pain VAS, 0 means no pain and 100 mm means extreme pain. For the gas VAS, 0 means no gas sensation and 100 mm means extreme gas sensation. The investigator measures the mark made by the participant in mm and records this for the value of either pain or gas.
Time Frame: Approximately 60 minutes after drug administration
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Pregabalin 75 mg | Pregabalin 200 mg | Placebo
Number analyzed (Participants) | 20 | 19 | 21
mm
  Sensation ratings for pain at 30 mm Hg | 47.4 (28.3) | 36.1 (28.4) | 46.0 (28.7)
  Sensation ratings for gas at 30 mm Hg | 53.4 (27.9) | 33.2 (19.6) | 46.6 (22.3)

3. Primary Outcome: Colonic Compliance
Description: Colonic compliance is a measure of the "stiffness" of the colon, that is, what pressure was needed to reach half the maximum value of the colon. After the barostat balloon catheter was inserted in the mid-descending or junction of the sigmoid and descending colon, the balloon was inflated. After an initial conditioning distension to 20 mm Hg, colonic compliance was measured by step-wise inflation with increments of 4 mm Hg. Colonic compliance was analyzed by a validated linear interpolation method. The pressure at half maximum volume serves as a summary of colonic compliance.
Time Frame: Approximately 60 minutes after drug administration
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Pregabalin 75 mg | Pregabalin 200 mg | Placebo
Number analyzed (Participants) | 20 | 19 | 21
mm Hg | 17.6 (5.1) | 19.1 (4.6) | 17.4 (4.8)

4. Primary Outcome: Postprandial Colonic Tone [Reported] as the Symmetric Percent [Change]in Baseline Colonic Barostat Balloon Volume
Description: The symmetric percent reduction in baseline colonic barostat balloon volume during the first 30 minutes postprandially (PP) corrected for the preprandial (30 min) tone, (symmetric percent change= 100*log_e[fasting/PP]). A positive symmetric percent change reflects a decrease in barostat balloon volume indicating a reduction in colonic tone. (The balloon was placed in the mid-descending or junction of the sigmoid and descending colon.)
Time Frame: The first 30 minutes postprandially, and preprandial (30 minutes)
Measure: Mean (Standard Deviation); unit: Symmetric percentage change
Arm/Group | Pregabalin 75 mg | Pregabalin 200 mg | Placebo
Number analyzed (Participants) | 20 | 19 | 21
Symmetric percentage change | 21.9 (12.4) | 35.3 (25.2) | 27.8 (21.8)

5. Primary Outcome: Postprandial Motility Index Over 30 Minutes
Description: The first 30 minute postprandial motility index (MI), MI = log_e [(number of contractions * sum of amplitudes)+1]
Time Frame: 30 minutes after the meal
Measure: Mean (Standard Deviation); unit: log mm Hg
Arm/Group | Pregabalin 75 mg | Pregabalin 200 mg | Placebo
Number analyzed (Participants) | 20 | 19 | 21
log mm Hg
  Motility index proximal colon at 30 minutes | 11.264 (1.609) | 11.764 (1.357) | 11.465 (1.339)
  Motility index distal colon at 30 minutes | 8.806 (3.095) | 9.783 (2.849) | 9.879 (2.235)

6. Secondary Outcome: Sensory Threshold for Gas
Description: The sensory threshold for first perception of gas was measured by stepwise inflation of the balloon in increments of 4 mm Hg at 60 second intervals. (The balloon was placed in the mid-descending or junction of the sigmoid and descending colon.) During this assessment participants were asked to report when they had the first perception of gas. The investigator recorded the threshold pressure at which the participants reported this sensation.
Time Frame: Approximately 60 minutes after drug administration
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Pregabalin 75 mg | Pregabalin 200 mg | Placebo
Number analyzed (Participants) | 20 | 19 | 21
mm Hg | 27.6 (18.3) | 34.3 (11.1) | 34.5 (16.8)

7. Secondary Outcome: Sensation Ratings for Pain at 16, 24, and 36 mm Hg Distension
Description: The mm Hg distensions refer to the barostat balloon, which was placed in the mid-descending or junction of the sigmoid and descending colon. Pain sensation was measured by a 100 mm long Visual Analog Scale (VAS). The VAS does not have any pre-set marks between the extremes. For the pain VAS, 0 means no pain and 100 mm means extreme pain. The investigator measures the mark made by the participant in mm and records this for the value of pain.
Time Frame: Approximately 60 minutes after drug administration
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Pregabalin 75 mg | Pregabalin 200 mg | Placebo
Number analyzed (Participants) | 20 | 19 | 21
mm
  Sensation ratings of pain at 16 mm distension | 28.70 (24.27) | 29.00 (28.47) | 34.29 (28.24)
  Sensation ratings of pain at 24 mm distension | 43.00 (30.66) | 36.84 (28.55) | 39.48 (29.78)
  Sensation ratings of pain at 36 mm distension | 44.30 (23.96) | 43.37 (26.94) | 47.62 (30.45)

8. Secondary Outcome: Sensation Ratings for Gas at 16, 24, and 36 mm Hg Distension
Description: The mm Hg distensions refer to the barostat balloon, which was placed in the mid-descending or junction of the sigmoid and descending colon. Gas sensation was measured by a 100 mm long Visual Analog Scale (VAS). The VAS does not have any pre-set marks between the extremes. For the gas VAS, 0 means no gas sensation and 100 mm means extreme gas sensation. The investigator measures the mark made by the participant in mm and records this for the value of either pain or gas.
Time Frame: Approximately 60 minutes after drug administration
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Pregabalin 75 mg | Pregabalin 200 mg | Placebo
Number analyzed (Participants) | 20 | 19 | 21
mm
  Sensation Ratings for Gas at 16 mm Hg distention | 37.40 (25.10) | 30.00 (25.25) | 37.14 (22.62)
  Sensation Ratings for Gas at 24 mm Hg distention | 44.05 (26.51) | 32.00 (21.83) | 42.76 (23.87)
  Sensation Ratings for Gas at 36 mm Hg distention | 49.65 (25.06) | 36.58 (22.42) | 46.24 (22.36)

9. Secondary Outcome: Gas Sensation Rating Averaged Across 4 Distension Pressures (16, 24, 30, and 36 mg Hg)
Description: The mm Hg distensions refer to the barostat balloon, which was placed in the mid-descending or junction of the sigmoid and descending colon. Gas sensation was measured by a 100 mm long Visual Analog Scale (VAS). The VAS does not have any pre-set marks between the extremes. For the gas VAS, 0 means no gas sensation and 100 mm means extreme gas sensation. The investigator measures the mark made by the participant in mm and records this for the value of gas. The values across the 4 distension pressures were averaged for this outcome measure.
Time Frame: Approximately 60 minutes after drug administration
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Pregabalin 75 mg | Pregabalin 200 mg | Placebo
Number analyzed (Participants) | 20 | 19 | 21
mm | 43.379 (23.413) | 33.391 (22.106) | 41.789 (22.278)
Statistical Analysis 1: Comparison: Pregabalin 75 mg vs Pregabalin 200 mg vs Placebo; ANCOVA for overall treatment effects; Test type: Superiority or Other; p = 0.14, ANCOVA — P-value not adjusted for multiple comparisons; alpha level of 0.05 used; mean value for 200 mg Pregabalin = 33.391, Standard Deviation 22.106 — A confidence interval was not calculated

10. Secondary Outcome: Pain Sensation Rating Averaged Across 4 Distension Pressures (16, 24, 30, and 36 mg Hg)
Description: The mm Hg distensions refer to the barostat balloon, which was placed in the mid-descending or junction of the sigmoid and descending colon. Pain sensation was measured by a 100 mm long Visual Analog Scale (VAS). The VAS does not have any pre-set marks between the extremes. For the pain VAS, 0 means no pain and 100 mm means extreme pain. The investigator measures the mark made by the participant in mm and records this for the value of pain. The values across the 4 distension pressures were averaged for this outcome measure.
Time Frame: Approximately 60 minutes after drug administration
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Pregabalin 75 mg | Pregabalin 200 mg | Placebo
Number analyzed (Participants) | 20 | 19 | 21
mm | 44.364 (23.478) | 35.301 (22.295) | 43.286 (23.678)
Statistical Analysis 1: Comparison: Pregabalin 75 mg vs Pregabalin 200 mg vs Placebo; ANCOVA for overall treatment effects; Test type: Superiority or Other; p = 0.12, ANCOVA — P-value not adjusted for multiple comparisons; alpha level of 0.05 used; mean value for 200 mg Pregabalin = 35.301, Standard Deviation 22.295 — A confidence interval was not calculated

ADVERSE EVENTS:
Time Frame: 5 hours after tube placement
Arm/Group | Pregabalin 75 mg | Pregabalin 200 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 14/20 | 19/19 | 9/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin 75 mg (N=20) | Pregabalin 200 mg (N=19) | Placebo (N=21)
Tachycardia (Cardiac disorders) | 9 (9) | 7 (7) | 8 (8)
Drowsiness (Nervous system disorders) | 4 (4) | 7 (7) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 7 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No